CLINICAL TRIAL: NCT06226649
Title: A Randomized Controlled Feasibility Trial Evaluating the Implementation of Digital Dyadic Empowerment Program (DDEP) on Lifestyle Modification for Chronic Kidney Disease Management
Brief Title: DDEP for Lifestyle Modification in Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Principal Investigator, Miaofen Yen, Professor, Department of Nursing, College of Medicine, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NHRI-EX113-11106PI
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Results first posted 2025-04-09 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Diseases
Keywords: feasibility studies; digital health; healthy lifestyle
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Dyadic Empowerment (Experimental): The intervention group (Digital Dyadic Empowerment) will utilize LINE, a prominent instant messaging App in Taiwan, to assist in lifestyle modification, along with support from the significant other.
  Interventions: Behavioral: Digital Dyadic Empowerment
- Control group (No Intervention): The control group receives routine education and care.

INTERVENTIONS:
Behavioral: Digital Dyadic Empowerment — The Digital Dyadic Empowerment Intervention utilizes LINE, a prominent instant messaging App in Taiwan, integrated with an extended application to deliver comprehensive lifestyle modification support to Chronic Kidney Disease (CKD) dyads. Key features of this intervention include:
  1. Access to CKD Health Education Information;
  2. Supportive Information for Significant Others;
  3. Physiological Values Logging for Self-Monitoring;
  4. Reminders for Clinical Appointments and Daily Self-Management Tasks;
  5. Kidney Health Diary for Lifestyle Modification Progress Tracking;
  6. Frequently Asked Questions (FAQs) and Consultation with Healthcare Providers.
  This intervention aims to enhance the overall well-being of CKD dyads by promoting education, self-monitoring, adherence to appointments, and efficient communication with healthcare providers.
  Other Names: LINE Official Account - Kidney Lifestyle
  Arms: Digital Dyadic Empowerment

SUMMARY:
This is a randomized controlled feasibility trial conducted on patients with Chronic Kidney Disease (CKD) and their significant other

DETAILED DESCRIPTION:
The trial will be conducted on 60 dyads, each comprising a CKD patient and a significant other, who will be randomly assigned into two groups. The intervention group will receive the Digital Dyadic Empowerment Program (DDEP) while the control group will receive routine education and care.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a diagnosis of Chronic Kidney Disease for at least six months;
2. The patient can identify a helpful significant other and both parties are willing to participate;
3. The patient can communicate in Mandarin or Taiwanese.

Exclusion Criteria:

1. The significant other is a healthcare provider;
2. The patient or the significant other has a mental illness diagnosis;
3. The patient is currently receiving renal replacement therapies.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miaofen Yen, PhD, Principal Investigator — National Cheng Kung University
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The "Enrollment" number (i.e., 120) in the Study Design Section reflects the total number of *participants* enrolled, and the number "Started" (i.e., 60) in the Participant Flow reflects the number of *dyads* assigned to Arms/Groups.
Groups:
- Digital Dyadic Empowerment: The intervention group (Digital Dyadic Empowerment) will utilize LINE, a prominent instant messaging App in Taiwan, to assist in lifestyle modification, along with support from the significant other.
  Digital Dyadic Empowerment: The Digital Dyadic Empowerment Intervention utilizes LINE, a prominent instant messaging App in Taiwan, integrated with an extended application to deliver comprehensive lifestyle modification support to Chronic Kidney Disease (CKD) dyads. Key features of this intervention include:
  1. Access to CKD Health Education Information;
  2. Supportive Information for Significant Others;
  3. Physiological Values Logging for Self-Monitoring;
  4. Reminders for Clinical Appointments and Daily Self-Management Tasks;
  5. Kidney Health Diary for Lifestyle Modification Progress Tracking;
  6. Frequently Asked Questions (FAQs) and Consultation with Healthcare Providers.
  This intervention aims to enhance the overall well-being of CKD dyads by promoting education, self-monitoring, adherence to appointments, and efficient communication with healthcare providers.
Period: Overall Study
Arm/Group | Digital Dyadic Empowerment | Control Group
Started | 30 (30 dyads (i.e., 30 patients and their 30 significant others) were randomly allocated to the intervention group.) | 30 (30 dyads (i.e., 30 patients and their 30 significant others) were randomly allocated to the control group.)
Completed | 26 | 29
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 4 | 1

BASELINE CHARACTERISTICS:
Population: Baseline data were not collected for those participants who dropped out of the study. Specifically, 4 dyads + 1 significant other in the intervention group and 1 dyad in the control group dropped out. As a result, there are 51 ([30-4]*2-1) participants from the intervention group and 58 ([30-1]*2) participants from the control group for baseline assessment. The overall number of baseline participants is therefore 109.
Groups:
- Total: Total of all reporting groups
Arm/Group | Digital Dyadic Empowerment | Control Group | Total
Number analyzed (Participants) | 51 | 58 | 109
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All 109 participants completed the baseline measure of Age. However, the age of the significant other or averaging the age of each dyad is not of great interest to our study and could be misleading as the role of the significant other (e.g., the patient's spouse, child, or grandchild) is not taken into account. Therefore, this measure reported here includes patient only to reflect the distribution of patient's age.
  years
    Patient: number analyzed (Participants) | 26 | 29 | 55
    Patient | 68.69 (10.45) | 68.76 (14.26) | 68.73 (12.49)
    Significant other: number analyzed (Participants) | 25 | 29 | 54
    Significant other | 51.56 (14.51) | 55.83 (15.82) | 53.85 (15.24)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All 109 participants completed the baseline measure of Sex. However, the count of sex for significant others or all participants together is not of great interest to our study and could be misleading as the role of the significant other (e.g., the patient's spouse, child, or grandchild) is not taken into account. Therefore, this measure reported here includes patient only.
  Participants
    Patient: number analyzed (Participants) | 26 | 29 | 55
    Patient: Female | 13 | 9 | 22
    Patient: Male | 13 | 20 | 33
    Significant other: number analyzed (Participants) | 25 | 29 | 54
    Significant other: Female | 16 | 22 | 38
    Significant other: Male | 9 | 7 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 51 | 58 | 109
eGFR [Mean (Standard Deviation); unit: ml/min/1.73m^2] — Estimated Glomerular Filtration Rate (eGFR) by the IDMS-MDRD Equation Population: This measure includes patient only.
  ml/min/1.73m^2
    number analyzed (Participants) | 26 | 29 | 55
    (all) | 46.29 (21.65) | 45.43 (29.79) | 45.84 (26.03)
CKD Stage [Count of Participants; unit: Participants] — A patient's stage of chronic kidney disease (CKD) based on eGFR. Criteria: Stage 1 (eGFR 90 or above), Stage 2 (eGFR 60-89), Stage 3a (eGFR 45-59), Stage 3b (eGFR 30-44), Stage 4 (eGFR 15-29), Stage 5 (eGFR less than 15). Higher stages (Stage 3b, Stage 4, and Stage 5) represent more advanced and severe progression of chronic kidney disease, with Stage 5 being the most advanced stage. Population: This measure includes patient only.
  Participants
    number analyzed (Participants) | 26 | 29 | 55
    Stage 1 | 2 | 1 | 3
    Stage 2 | 4 | 7 | 11
    Stage 3a | 8 | 6 | 14
    Stage 3b | 5 | 4 | 9
    Stage 4 | 5 | 6 | 11
    Stage 5 | 2 | 5 | 7
TTM Stage [Number; unit: dyad] — The TTM stages of change in lifestyle modification were assessed using five statements based on the Transtheoretical Model (TTM). Patients and their significant others self-assessed their motivation for lifestyle modification, identifying as being in the "precontemplation," "contemplation," "preparation," "action," or "maintenance" stage. Population: This measure was reported jointly by the patient and the significant other within each dyad.
  dyad
    Precontemplation | 2 | 1 | 3
    Contemplation | 0 | 1 | 1
    Preparation | 5 | 1 | 6
    Action | 7 | 7 | 14
    Maintenance | 12 | 19 | 31
Health Promoting Lifestyle [Mean (Standard Deviation); unit: units on a scale] — Patients' lifestyles were assessed using the Chinese version of the Health Promoting Lifestyle Profile-II (HPLP-II), a validated scale with 52 items rated on a 4-point Likert scale. The total score ranges from 52 to 208, with higher scores indicating better health-promoting behavior. Population: This measure includes patients only.
  units on a scale
    number analyzed (Participants) | 26 | 29 | 55
    (all) | 142.19 (24.8) | 140.69 (21.7) | 141.40 (23.04)
Adherence to Healthy Behaviors [Mean (Standard Deviation); unit: units on a scale] — Patients' adherence to healthy behaviors over the past month was measured using the Adherence to Healthy Behaviors Scale (AHBS). The scale includes 13 items rated on a 5-point Likert scale, with total scores ranging from 0 to 52. Higher scores indicate better adherence. Population: This measure includes patient only.
  units on a scale
    number analyzed (Participants) | 26 | 29 | 55
    (all) | 45.23 (6.0) | 44.97 (5.5) | 45.09 (5.7)
Helping Relationships from Significant Others [Mean (Standard Deviation); unit: units on a scale] — Patients' perceived support from their significant others over the past month was assessed using the Chinese version of the Helping Relationships from Significant Others Scale (HRSO). The scale consists of 15 items rated on a 7-point Likert scale, with total scores ranging from 15 to 105, with higher scores indicating better support. Population: This measure includes patient only.
  units on a scale
    number analyzed (Participants) | 26 | 29 | 55
    (all) | 88.58 (18.2) | 90.45 (12.0) | 89.56 (15.1)
Dyadic Adjustment [Mean (Standard Deviation); unit: units on a scale] — The quality of the relationship between the patient and their significant other was assessed using the 7-item Dyadic Adjustment Scale (DAS-7). The first six items are rated on a 6-point scale, while the seventh item is rated on a 7-point scale, with total scores ranging from 0 to 36. Higher scores indicate better relationship quality. Population: This scale was measured for both patients and their significant others. Specifically, 26 dyads from the intervention group and 29 dyads from the control group completed the baseline assessment for this scale. However, one significant other from the intervention did not complete the baseline assessment for this scale. As a result, 51 (26*2-1) participants from the intervention group and 58 (29*2) participants from the control group were included for the analysis population of this scale.
  units on a scale | 20.67 (6.13) | 21.60 (6.00) | 21.17 (6.05)
Quality of Life [Mean (Standard Deviation); unit: units on a scale] — The Taiwanese version of the World Health Organization Quality of Life Questionnaire (WHOQOL-BREF) was used to assess the quality of life of patients and their significant others over the past two weeks. The first item assessing general quality of life, rated on a 5-point Likert scale (score range: 1 to 5), was reported for this measure. Higher scores indicate better quality of life.
  units on a scale | 3.61 (0.70) | 3.60 (0.70) | 3.61 (0.69)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in eGFR at 3 Months (Patient-specific)
Description: For each patient, change from Baseline (Followup score - Baseline score) in the estimated Glomerular Filtration Rate (eGFR) by the IDMS-MDRD Equation at 3 months was obtained through the patient's biochemical test reports. Higher eGFR numbers generally indicate better kidney functions.
Time Frame: Before initial intervention and 3 months after initial intervention
Population: The test of eGFR was conducted only on patient participants.
Measure: Mean (95% Confidence Interval); unit: ml/min/1.73m^2
Arm/Group | Digital Dyadic Empowerment | Control Group
Number analyzed (Participants) | 26 | 29
ml/min/1.73m^2 | -1.71 [-3.58 to 0.17] | -4.12 [-9.11 to 0.86]

2. Primary Outcome: Change From Baseline in CKD Stage at 3 Months (Patient-specific)
Description: For each patient, the change from Baseline in CKD stage at 3 months was obtained by comparing the CKD stage at baseline and at follow-up, converted into the following three categories: (1) recover (e.g., from Stage 3a [at baseline] to Stage 2 [at follow-up]); (2) stable (e.g., remaining Stage 3a at both baseline and follow-up); and (3) progress (e.g., from Stage 3a [at baseline] to Stage 3b [at follow-up]).
Time Frame: Before initial intervention and 3 months after initial intervention
Population: This measure was conducted only on the patient participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Dyadic Empowerment | Control Group
Number analyzed (Participants) | 26 | 29
Participants
  Recover | 2 | 4
  Stable | 18 | 20
  Progress | 6 | 5

3. Primary Outcome: Change From Baseline in TTM Stage at 3 Months
Description: For each dyad, change from Baseline in TTM stage at 3 months was obtained by comparing the TTM stage of change at baseline and at follow-up, converted into the following three categories: (1) regress (e.g., from Preparation [at baseline] to Contemplation [at follow-up]); (2) maintain (e.g., remaining Action at both baseline and follow-up); and (3) advance (e.g., from Action [at baseline] to Maintanece [at follow-up]).
Time Frame: Before initial intervention and 3 months after initial intervention
Population: This measure was reported jointly by the patient and the significant other within each dyad.
Measure: Number; unit: dyad
Arm/Group | Digital Dyadic Empowerment | Control Group
Number analyzed (Participants) | 51 | 58
dyad
  Regress | 4 | 5
  Maintain | 14 | 19
  Advance | 8 | 5

4. Primary Outcome: Change From Baseline in Health Promoting Lifestyle at 3 Months (Patient-specific)
Description: For each patient, change from Baseline (Followup score - Baseline score) in patient's Health Promoting Lifestyle at 3 months was assessed using the Chinese version of the Health Promoting Lifestyle Profile-II (HPLP-II), a validated scale with 52 items rated on a 4-point Likert scale. The total scores range from 52 to 208, with higher scores indicate better health-promoting behavior.
Time Frame: Before initial intervention and 3 months after initial intervention
Population: This questionnaire was only administrated to the patient participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Digital Dyadic Empowerment | Control Group
Number analyzed (Participants) | 26 | 29
score on a scale | 5.96 [-0.77 to 12.70] | -8.17 [-18.52 to 2.18]

5. Primary Outcome: Change From Baseline in Quality of Life at 3 Months
Description: For each participant, change from Baseline (Followup score - Baseline score) in Quality of Life at 3 months was assessed using the first item of the Taiwanese version of the World Health Organization Quality of Life Questionnaire (WHOQOL-BREF). The item was rated on a 5-point Likert scale, ranging from 1 to 5. Higher scores indicate better quality of life.
Time Frame: Before initial intervention and 3 months after initial intervention
Population: This scale was measured for both patients and their significant others. Specifically, 26 dyads from the intervention group and 29 dyads from the control group completed the baseline assessment for this scale. However, one significant other from the intervention did not complete the baseline assessment for this scale. As a result, 51 (26*2-1) participants from the intervention group and 58 (29*2) participants from the control group were included for the analysis population of this scale.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Digital Dyadic Empowerment | Control Group
Number analyzed (Participants) | 51 | 58
units on a scale | -0.02 [-0.21 to 0.17] | -0.16 [-0.40 to 0.09]

6. Secondary Outcome: Change From Baseline in Adherence to Health Behaviors at 3 Months (Patient-specific)
Description: For each patient, change from Baseline (Followup score - Baseline score) in patient's adherence to healthy behaviors was measured using the Adherence to Healthy Behaviors Scale (AHBS). The scale includes 13 items rated on a 5-point Likert scale, with total scores ranging from 0 to 52. Higher scores indicate better adherence.
Time Frame: Before initial intervention and 3 months after initial intervention
Population: This questionnaire was only administrated to the patient participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Digital Dyadic Empowerment | Control Group
Number analyzed (Participants) | 26 | 29
score on a scale | 1.81 [0.17 to 3.45] | 0.10 [-2.33 to 2.54]

7. Secondary Outcome: Change From Baseline in Helping Relationships From Significant Others at 3 Months (Patient-specific)
Description: For each patient, change from Baseline (Followup score - Baseline score) in patient's Helping Relationships from Significant Others at 3 months was assessed using the Chinese version of the Helping Relationships from Significant Others Scale (HRSO).The scale consists of 15 items rated on a 7-point Likert scale, with total scores ranging from 15 to 105. Higher scores indicate better support from the significant other.
Time Frame: Before initial intervention and 3 months after initial intervention
Population: This questionnaire was only administrated to the patient participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Digital Dyadic Empowerment | Control Group
Number analyzed (Participants) | 26 | 29
score on a scale | 4.42 [-0.90 to 9.75] | -8.86 [-15.34 to -2.39]

8. Secondary Outcome: Change From Baseline in Dyadic Adjustment at 3 Months
Description: For each participant, change from Baseline (Followup score - Baseline score) in Dyadic Adjustment at 3 months was assessed using the 7-item Dyadic Adjustment Scale (DAS-7). The first six items are rated on a 6-point scale, while the seventh item is rated on a 7-point scale. The total scores range from 0 to 36, with higher scores indicating better relationship quality.
Time Frame: Before initial intervention and 3 months after initial intervention
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Digital Dyadic Empowerment | Control Group
Number analyzed (Participants) | 51 | 58
score on a scale | 2.49 [0.15 to 4.83] | -1.47 [-3.12 to 0.19]

ADVERSE EVENTS:
Time Frame: 9 months
Description: For this study, adverse events are defined as any discomfort reported by all participants from using the DDEP platform for the intervention group, or from completing questionnaires for all participants for both the intervention or the control groups.
Arm/Group | Digital Dyadic Empowerment | Control Group
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

LIMITATIONS AND CAVEATS:
Since this is a feasibility trial, the change from baseline estimates for all outcomes were underpowered, and therefore 95% confidence intervals (CIs) were reported instead.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-04): https://cdn.clinicaltrials.gov/large-docs/49/NCT06226649/Prot_SAP_000.pdf